CLINICAL TRIAL: NCT06613958
Title: Older Adults Exercising On Time
Acronym: ON TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Organisation of Scientific Research (NWO) (Unknown); Centre for Human Drug Research, Netherlands (Other); Chrono@Work (Unknown); Corsano Health B.V. (Industry); M-Path Leuven (Unknown)
Responsible Party: Principal Investigator, dvanheemst, Principal investigator, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL82335.058.22
Record Dates: First submitted 2024-03-12; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Insomnia; Circadian Rhythm Disorders
Keywords: Chronoactivity; Sleep; Circadian rhythm; Exercise timing
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronobiology Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will perform a randomized two-armed cross-over study. Both groups will start with the sedentary period. Depending on the intervention arm, participants will then undergo the active morning intervention or active evening intervention first, followed by the other intervention. There will be a total of two washout periods both lasting 7 days, one between the sedentary period and first intervention and one between the first and second intervention to prevent or minimize 'carry over' of previous intervention effect. The two interventions and the sedentary period will last 14 days each and contain a 'calibration period' (7 days) and a 'measurement week' (7 days). The total study duration will be 8 weeks and the study will largely take place at the participants' home except for the training sessions (Vitality Clubs) that will take place at an outdoor sports facility in the municipality of Leiden and the study site visits which will take place in the LUMC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Order of interventions: Sedentary - Active morning - Active Evening
  Interventions: Behavioral: Physical activity timing
- Group 2 (Other): Order of the interventions: Sedentary - Active Evening - Active Morning
  Interventions: Behavioral: Physical activity timing

INTERVENTIONS:
Behavioral: Physical activity timing — The investigators will compare our interventions to a 14-day period of sedentary behavior, during which the participant will refrain from any moderate to vigorous exercise. Next, participants will participate in two interventions consisting each of a 14-day physical activity regimen. The active morning and active evening interventions are equal in content. Both groups will be instructed to refrain from any moderate to vigorous exercise for the rest of the day. Per intervention, a total of eight Vitality Club training session comprising of a combination of aerobic endurance training and resistance exercise training will be given by a trained sports coach or physical therapist specialized in geriatric physical therapy. During the weekends, participants will be asked to perform a 'relative rest' session with some light activity during the training time window of the intervention arm.
  Other Names: Active morning (exercise program from 10:00 - 11:00 in the morning); Active evening (exercise program from 19:30 - 20:30 in the evening); Sedentary period (no exercise)

SUMMARY:
There are indications from epidemiological cohort studies and animal experiments that timing of physical activity (also referred as "chronoactivity"), irrespective of intensity, impacts health and disease. In view of the detrimental effects of circadian misalignment, the large group of older people suffering from sleep problems, and the seeming importance of chronoactivity, the investigators will perform a randomised cross-over study that aims to uncover the effect of timing of physical activity on insomnia severity and related(circadian) health parameters in older adults with self-reported sleep problems. Here, the investigators hypothesize that timing of physical activity has a beneficial impact on insomnia symptoms and on circadian rhythms of additional health parameters (e.g., metabolic, psychosocial) in older people. To study this research hypothesis, the investigators will examine the effect of physical activity timing on insomnia severity in older adults with self-reported sleep problems. In addition, the investigators will examine the effect of physical activity timing on exploratory rhythmic parameters of biological clock function, physiology and metabolism, mental health, behavioural factors, and immune and cell signalling functions. For this study, a two-armed randomised cross-over study, Dutch speaking older adults between 60 and 80 years old (male and female) and having sleep problems (insomnia severity index>10 points) from the general population in the Netherlands will be selected as participants for this study. Participants will perform one sedentary period and two period of increased physical activity with different daily patterns: 1)active morning; 2) active evening with a duration of 14 days each. In both active intervention arms, participants will follow an exercise program containing outdoor physical exercise sessions (Vitality Club) containing endurance and strength exercises, relative rest days of 30 minutes light intensity physical activity, and one Active@Home program; a 1-hour training session of various moderate to vigorous activities. The training sessions will be held either in the morning or evening (depending on the intervention arm) and will be one hour long. Study outcomes will be compared between the different intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 and 80 years old
* Retired
* Long lasting sleep problems (as assessed by a the screening questionnaire administered telephonically and by the ISI which will be filled out during the screening visit)
* Access to and ability to use a smart phone (Android or Apple)

Exclusion Criteria:

* Currently employed or working
* Extreme sleep chronotypes (measured by the Munich chronotype questionnaire)
* Participation in any sort of fasting regimen (e.g. intermitted fasting or Ramadan)
* Experienced recent (<6 months) adverse life events (e.g., death of partner)
* Abnormal values in glucose metabolism, thyroid, liver or kidney function, or inflammation markers that after examination of the study doctor need immediate attention of a general practitioner or specialist.
* Diagnosed clinical depression
* Diagnosed neurodegenerative diseases (e.g. dementia or Parkinson's disease)
* Diagnosed sleep apnoea
* Diagnosed restless legs syndrome
* Use of beta-adrenergic blocking agents
* Use of sleep medication*
* Injuries or other severe physical conditions (such as active arthrosis) that inhibits physical activity
* Travelled across time zones one week prior to start of study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | 4 times in total: at baseline T-3 (T= week), at T2 , T5, and at T8 (endline).
  Score on Insomnia Severity Index (ISI). Participants will be asked to fill out the ISI questionnaire (Dutch version) The ISI questionnaire consists of 7 questions and outcomes include: 'No clinically significant insomnia (0-7 points)', 'Subthreshold insomnia (8-14 points)', 'Moderate severity clinical insomnia (15-21 point), and 'Severe clinical insomnia (22-28 points)'.

SECONDARY OUTCOMES:
Dim light melatonin onset (DLMO) | 3 times in total: two weeks, five weeks and eight weeks after baseline.
  Participants will be asked to perform/collect 7 buccal swabs in a time range of 5 hours prior to bedtime to 1 hour after bedtime to measure the melatonin pattern DLMO one evening at the end of each intervention. This measurement will be done according to the standard protocol from Chrono@Work (Groningen, The Netherlands) in dim light conditions. Participants will be carefully instructed beforehand on the procedure. Melatonin levels will be shown in Pg/ml
Ecological monitoring assessment | 3 periods in total of one week each: the second week, the fifth week and the eighth week.
  During the measurement week, participants will be asked to fill out the eEMA questionnaire in the Leuven mPath app 4 times a day on set times (between 7-9 AM, 12-2 PM, 4-6 PM and 8-10 PM). Participants will receive a pop-up on their smartphones and will have a window of 2 hours to fill in the questionnaire. The questionnaire consists of multiple questions that gather information on current mood/feelings divided into multiple dimensions: positive affectivity, negative affectivity, energetic arousal and cognition. A visual analogue scale will be used to answer the questions. To minimize the burden of this repeated questionnaire, the time needed to fill out the questionnaire is limited to approximately 3 minutes.
Sleep quality - sleep duration | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Objective sleep quality will be monitored with the Withings Sleep Analyzer (Withings, Issy-les-Moulineaux, France) . Prior to the study, the Withings Sleep Analyzer will be installed in the participants bed. A smart phone is required to set-up the device and the devices must be connected to a Wi-Fi to be able to send data to the cloud. After set-up no link to the smartphone is required. The device must be connected to power.
  Sleep duration, pattern of and duration spent in different sleep stages (deep, REM, and light sleep), sleep latency, sleep efficiency, and sleep regularity.
Sleep quality - sleep latency | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Objective sleep quality will be monitored with the Withings Sleep Analyzer (Withings, Issy-les-Moulineaux, France) . Prior to the study, the Withings Sleep Analyzer will be installed in the participants bed. A smart phone is required to set-up the device and the devices must be connected to a Wi-Fi to be able to send data to the cloud. After set-up no link to the smartphone is required. The device must be connected to power.
  Sleep duration, pattern of and duration spent in different sleep stages (deep, REM, and light sleep), sleep latency, sleep efficiency, and sleep regularity.
Sleep quality - sleep stages | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Objective sleep quality will be monitored with the Withings Sleep Analyzer (Withings, Issy-les-Moulineaux, France) . Prior to the study, the Withings Sleep Analyzer will be installed in the participants bed. A smart phone is required to set-up the device and the devices must be connected to a Wi-Fi to be able to send data to the cloud. After set-up no link to the smartphone is required. The device must be connected to power.
  Sleep duration, pattern of and duration spent in different sleep stages (deep, REM, and light sleep), sleep latency, sleep efficiency, and sleep regularity.
Sleep quality - sleep efficiency | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Objective sleep quality will be monitored with the Withings Sleep Analyzer (Withings, Issy-les-Moulineaux, France) . Prior to the study, the Withings Sleep Analyzer will be installed in the participants bed. A smart phone is required to set-up the device and the devices must be connected to a Wi-Fi to be able to send data to the cloud. After set-up no link to the smartphone is required. The device must be connected to power.
  Sleep duration, pattern of and duration spent in different sleep stages (deep, REM, and light sleep), sleep latency, sleep efficiency, and sleep regularity.
Sleep quality - sleep regularity | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Objective sleep quality will be monitored with the Withings Sleep Analyzer (Withings, Issy-les-Moulineaux, France) . Prior to the study, the Withings Sleep Analyzer will be installed in the participants bed. A smart phone is required to set-up the device and the devices must be connected to a Wi-Fi to be able to send data to the cloud. After set-up no link to the smartphone is required. The device must be connected to power.
  Sleep duration, pattern of and duration spent in different sleep stages (deep, REM, and light sleep), sleep latency, sleep efficiency, and sleep regularity.
Biological assessment: clock gene expression | 4 times in total: at baseline (3 weeks before start of the study), at the second , fifth, and eighth week
  Paxgene 1x 2.5 ml 7,5 ml RNA Gene expression clock genes (in batch)
Biological assessment: metabolomics | 4 times in total: at baseline (3 weeks before start of the study), at the second , fifth, and eighth week
  EDTA 1x 2 ml 6 ml plasma Metabolomics (in batch)
Biological assessment: proteomics | 4 times in total: at baseline (3 weeks before start of the study), at the second , fifth, and eighth week
  EDTA 1x 2 ml 6 ml plasma proteomics (in batch)
Biological assessment: glucose metabolism | 4 times in total: at baseline (3 weeks before start of the study), at the second , fifth, and eighth week
  EDTA 1x 2 ml 2 ml plasma HbA1c, Insulin, glucose,
Biological assessment: biomarkers for inflammation, thyroid, kidney and liver function | 4 times in total: at baseline (3 weeks before start of the study), at the second , fifth, and eighth week
  Serum 1x 3.5 ml 14 ml serum eGRF/creatinin, Hs-CRP, Gamma GT, ASAT, ALAT, TSH, ft4 (in batch)
Food capturing | 3 periods in total of one week each: week two, week five, and at week eight.
  Participants will log their daily food intake during each measurement week by using a food diary that will be distributed prior to the start of the study. Frequency and timing of food intake will be assessed.
Heart rate | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Participants will wear the Corsano Cardiowatch 287-2 (Corsano Health, The Hague, the Netherlands) wrist band on their right wrist continuously during the study period. The wristband is multifunctional and is waterproof. Participants will wear the wrist band 24 hours a day. The HR is measured using a PPG (photoplethysmogram, i.e., optically obtained volumetric measurement) and ECG. The manufacturer supplies the algorithm for converting the PPG/ECG signals into a set of HR values. All data from the Cardiowatch is available real time and is transferred from the watch to the smartphone using a clinical trial app, developed by the provider, which allows the researcher to retrieve live vital sign data while conducting a blinded study.
Heart rate variability | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Participants will wear the Corsano Cardiowatch 287-2 (Corsano Health, The Hague, the Netherlands) wrist band on their right wrist continuously during the study period. The wristband is multifunctional and is waterproof. Participants will wear the wrist band 24 hours a day. The HR is measured using a PPG (photoplethysmogram, i.e., optically obtained volumetric measurement) and ECG. The manufacturer supplies the algorithm for converting the PPG/ECG signals into a set of HR values. All data from the Cardiowatch is available real time and is transferred from the watch to the smartphone using a clinical trial app, developed by the provider, which allows the researcher to retrieve live vital sign data while conducting a blinded study.
Core body temperature | 3 periods in total of 2 weeks each: weeks 1-2 , weeks 4-5, and weeks 7-8.
  Core body temperature will be continuously measured by the Cardiowatch 287-2 in degrees Celcius. This parameter will be derived through an algorhythm of combined data from Heatflux sensor and PPG signal. Diurnal patterns of core body temperature as well as the time of lowest daily temperature will be derived from this data.

CONTACTS AND LOCATIONS:
Overall Officials: Diana van Heemst, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT06613958/Prot_SAP_000.pdf